CLINICAL TRIAL: NCT04367688
Title: Delivery of Pre-exposure Prophylaxis to Individuals With High Sexual Risk of HIV Infection in Hong Kong - an Implementation Study
Brief Title: HIV Pre-exposure Prophylaxis Implementation Hong Kong Study
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shui-Shan Lee, MD, Professor, Chinese University of Hong Kong
Other Study IDs: MSS325R
Record Dates: First submitted 2020-04-26; First posted 2020-04-29 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: HIV Infections
Keywords: HIV; pre-exposure prophylaxis; adherence; antiretroviral
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Emtricitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate 300 mg / emtricitabine 200 mg — daily use for PrEP

SUMMARY:
While pre-exposure prophylaxis (PrEP) is widely recommended and a number of pilot studies are on-going worldwide, progress of its implementation in the real world setting has been slow, especially in Asia. This study aims to develop a service model for PrEP delivery and test its operability in the real world setting. In this implementation study, 400 individuals with high sexual risk of HIV infection who fulfil eligibility criteria would be recruited. Eligible participants would receive one year of daily tenofovir disoproxil fumarate 300mg / emtricitabine 200mg (TDF/FTC) for free. A client-initiated approach would be adopted, requiring participants to self-arrange for regular HIV/sexually transmitted infections (STI) testing. An online system would be developed to facilitate participants to plan for testing and consultation for accessing PrEP. Questionnaire at baseline and subsequent monthly follow-up would be administered to assess behaviour, monitor adverse effects and drug adherence, the latter coupled with the completion of an online diary. Testing of HIV and creatinine would be performed using point-of-care test or by phlebotomy during clinical visits. Blood samples would be collected for archiving. Around 40 participants would be invited to join an in-depth interview in the later part of the study to evaluate the service model. The main outcome measures are: PrEP service adherence, PrEP drug adherence, prevalence of drug intolerance, prevalence of unprotected sex in the study period, incidence of HIV and STI

ELIGIBILITY:
Inclusion Criteria:

* Can communicate in written and spoken English or Chinese
* Is normally resident in Hong Kong
* Has tested HIV antibody negative in the past 3 months
* Has more than 1 episode of unprotected sex (especially anal sex) in the preceding 6 months
* Has any one of the following experiences in the past 6 months: chemsex engagement, group sex, multiple sex partners, STI diagnosis, having sex partner(s) with HIV+ve status
* Is inclined to engage in high risk sexual activities

Exclusion Criteria:

* Chronic HBV infection (HBsAg +ve)
* Impaired renal function, defined as estimated glomerular filtration rate (eGFR) < 60mL/min/1.73m2
* Having any form of mental illnesses
* Inability or refusal to give consent
* Prisoners or any institutionalised persons
* Pregnant or planning to get pregnant (for female)
* Injection drug user

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with high risk sexual behaviours for HIV transmission who are referred by government/public service or non-government service in Hong Kong or self-referred for enrolment in a PrEP program
Sampling Method: Non-Probability Sample
Enrollment: 339 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
adherence to PrEP service | 12 months
  attending the PrEP service with prescription and HIV tests regularly in accordance with protocol
adherence to PrEP regimen | 12 months
  proportion adherent to daily TDF/FTC

CONTACTS AND LOCATIONS:
Overall Officials: Shui Shan Lee, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No